CLINICAL TRIAL: NCT00516633
Title: Does Improved Information in the Form of Group Discussions With Parents of Newly Diagnosed Asth-Matic Children Lead to a Better Quality of Life for the Families, an Improved Adherence and Better Devel-Opment of the Lung Function of the Children?
Brief Title: Intervention Study to Improve Adherence in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Värmland County Council, Sweden (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIVFOU-8215
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Asthma
Keywords: Asthma; Adherence; Burden of asthma; Quality of life; Questionnaires
MeSH Terms: conditions — Asthma | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CG (No Intervention): The control group had regular individual information and support in connection with ordinary clinical follow-ups
- IG (Experimental): The intervention group had extra support and information in the form of four group discussions with parents
  Interventions: Behavioral: Extra information and support

INTERVENTIONS:
Behavioral: Extra information and support — Four group discussions with parents in close connection to diagnosing the children
  Arms: IG

SUMMARY:
We wanted to investigate if it was possible to improve adherence to prescriptions and advice in pre-school children with newly diagnosed asthma. The intervention was intense information and support in the form of four group discussions with the parents of four children in close connection to diagnosing the child. The control children received the usual care with individual polyclinic visits to the physi-cian/nurse. We evaluated the effect with the help of questionnaires, physical examinations, blood tests, lung function tests and control of treatment adherence after 18 months and 6 years.

DETAILED DESCRIPTION:
Poor adherence to the prescribed regimen of medication is one of the major obstacles to successful treatment of many chronic diseases, in the case of both grown-ups and children. In 1998 we initiated a randomized, prospective intervention study with per protocol design involving 60 young children re-cently diagnosed as having asthma and with a high risk that this condition would persist.

The parents of the children in the intervention group received extra support and information in the form of group discussions, whereas the control patients were treated in a routine manner. All children 0-6 years of age who fulfilled at least one of the criteria for risk of persistent asthma among the 9410 children in our catchments area were evaluated at our out-patient clinic during a period of 1.5 years beginning in 1998. Of the 66 patients thus identified the parents of 6 declined to participate and the remaining 60 children were randomized consecutively in groups of four by a nurse to either the inter-vention or the control group. The groups turned out to be well-matched.

All of the children received the usual management and care, including individual oral and written information concerning how to deal with their asthma. The intervention consisted of additional infor-mation and support in a group setting, with three 1.5-hour meetings soon after inclusion in the study (with 70% participation, no gender difference) and a fourth meeting 6 months later (with 40% partici-pation). The three nurses, three pediatricians and two psychologists who performed this investigation were also in charge of the intervention, i.e. the study was not blinded.

The initial examination included a clinical examination, spirometry, chest x-ray, examination of the patients' records and questionnaires concerning issues of adherence, burden of asthma and quality of life (Pediatric Caregiver's Quality of Life Questionnaire, PACQLQ). This Questionnaire was filled out separately by the fathers and the mothers and a change of > 0.5 units on a 7-point scale was considered to be clinically important. The blood and urine were analyzed for inflammatory parameters. Skin prick tests were performed being considered positive if the mean diameter of the wheal was >3 mm. The al-lergen extracts used were Soluprick® (ALK-Albello A/S, Denmark) and included egg, birch, timothy, mugwort, dog, cat, horse and Dermatophagoides pteronyssinus. RAST® testing (Pharmacia Diagnos-tics & Upjohn AB) with the same allergens (considered positive when the IgE-level was >0.7 kU/l) and Phadiatop® testing (Pharmacia Diagnostics & Upjohn AB) (considered positive if the value > 1.0 kU/l) were also performed.

The children made regular visits to their own pediatrician and nurse during the subsequent years and their medical records have been continuously updated and computerized. The examination after 6 years was performed during 2005. In this context each child was examined and interviewed, in the company of one or both parents and the examination being the same as earlier, except that no chest x-ray or objective assessment of adherence was carried out.

This time separate questionnaires addressed to the child (the Pediatric Asthma Quality of Life Questionnaire) and to the child and parent together (the Asthma Control Questionnaire) were included, with a value of < 0.75 considered as being an indicator of good asthma control. Furthermore exhaled NO was measured with the help of the NIOXMINO® Airway Inflammation Monitor (Aerocrine AB, Solna, Sweden), utilizing a 10-sec expiration at a constant flow rate of 0.05 l/s. In addition, we per-formed dry-air tests (Aiolos AB, Karlstad, Sweden), in connection with which a fall in FEV1 of > 10% was considered pathological.

During the follow-up parents and doctors estimated adherence on a visual analogue scale (VAS). The children were told to begin taking high doses of ICS (0.2 mgx4) as soon as they caught a cold, even before they had any asthmatic symptoms, and to subsequently reduce the dose gradually during the first week, stopping medication when they no longer had any symptoms. When symptoms of asthma developed they were instructed to continue ICS for one month and, if they had experienced three or more exacerbations during a12-month period, to continue this treatment for another six months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma and fullfilling the criteria utilized to indicate high risk for persistent asthma: the presence of atopic disease among close relatives, confirmed allergy, symptoms of another atopic disease or asthma that appeared between bouts of the common cold.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 1998-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Adherence | 18 months and 6 years

SECONDARY OUTCOMES:
Burden of asthma on the individual and on the health care system | 18 months and 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Hedlin, Professor, Study Chair — Karolinska Institutet
Locations (1):
- Barn-ungdomsmedicinska mottagningen VC Gripen, Karlstad, Sweden

REFERENCES:
- [Result] Hederos CA, Janson S, Hedlin G. Group discussions with parents have long-term positive effects on the management of asthma with good cost-benefit. Acta Paediatr. 2005 May;94(5):602-8. doi: 10.1111/j.1651-2227.2005.tb01946.x. PMID 16188750
- [Result] Hederos CA. Neuropsychologic changes and inhaled corticosteroids. J Allergy Clin Immunol. 2004 Aug;114(2):451-2. doi: 10.1016/j.jaci.2004.03.045. No abstract available. PMID 15341026
- [Result] Hederos CA, Janson S, Andersson H, Hedlin G. Chest X-ray investigation in newly discovered asthma. Pediatr Allergy Immunol. 2004 Apr;15(2):163-5. doi: 10.1046/j.1399-3038.2003.00098.x. PMID 15059194